CLINICAL TRIAL: NCT06165042
Title: Evaluation of Silver Diamine Fluoride Application in Molar-Incisor Hypomineralisation-Affected Molars
Brief Title: Silver Diamine Fluoride in Molar-Incisor Hypomineralisation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MarmaraPedo
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Molar-Incisor Hypomineralisation
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glass hybrid restorative system (Experimental): (Equia Forte, GC Europe, Leuven, Belgium)
  Interventions: Other: glass hybrid restorative system
- Fluoride varnish + Glass hybrid restorative (Experimental): Fluoride varnish (SDI Riva Star)+ Glass hybrid restorative (Equia Forte, GC Europe, Leuven, Belgium)
  Interventions: Other: Fluoride varnish + Glass hybrid restorative system

INTERVENTIONS:
Other: glass hybrid restorative system — In the teeth where the indication is identified, selective caries removal will be performed to eliminate the decayed tooth tissue. Subsequently, for each patient in the study apply glass hybrid restorative system (Equia Forte, GC Europe, Leuven, Belgium)
  Arms: Glass hybrid restorative system
Other: Fluoride varnish + Glass hybrid restorative system — In the teeth where the indication is identified, selective caries removal will be performed to eliminate the decayed tooth tissue. Subsequently, for each patient in the study apply Fluoride varnish (SDI Riva Star)+ Glass hybrid restorative (Equia Forte, GC Europe, Leuven, Belgium)
  Arms: Fluoride varnish + Glass hybrid restorative

SUMMARY:
The objective of this study is to assess the efficacy of silver diamine fluoride application in molars affected by molar-incisor hypomineralization. Additionally, the study aims to evaluate the effectiveness of the combined application of silver diamine fluoride, commonly used for dentin hypersensitivity, with a glass hybrid restorative system. The goal is to mitigate sensitivity and improve chewing functions in teeth affected by molar-incisor hypomineralization.

DETAILED DESCRIPTION:
In a research study focusing on 120 children aged 8-13 with molar incisor hypomineralization (MIH), a comprehensive examination of 240 teeth will be conducted. Study will employ selective caries removal to eliminate decay and subsequently apply restorations. The two intervention groups are delineated as follows:

Group 1: Glass hybrid restorative system (Equia Forte, GC Europe, Leuven, Belgium)

Group 2 : Restoration involving fluoride varnish (SDI Riva Star) + glass hybrid restorative system (Equia Forte, GC Europe, Leuven, Belgium)

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 8 and 13 who are cooperative, having at least 2 teeth with a BAKH-TII score of 4a or 4b.
* Complete occlusion of teeth with MIH.
* Presence of signs of pulpal pathology with symptoms in the teeth included in the study during the pre-treatment clinical examination (absence of spontaneous and prolonged pain, no percussion and palpation sensitivity, no swelling or fistula in soft tissue, presence of periapical radiolucency in radiographs, and absence of internal or external resorption).
* Additionally, no parafunctional habits (e.g., bruxism) and no malocclusion (posterior crossbite).
* Good general health condition, without systemic illnesses.
* Absence of silver allergy.

Exclusion Criteria:

* Non-cooperative individuals.
* Having MIH severity outside the specified scoring.
* Presence of systemic diseases.
* Lack of complete occlusion in the molars.
* Presence of parafunctional habits.
* Presence of pulpal pathology.
* Individuals with a silver allergy.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
United States Public Health Service (USPHS): Retention, marginal compliance and gingival health criteria | 1.5 -2 year
  Restorations were evaluated to determine success according to modified United States Public Health Service (USPHS) criteria for marginal adaptation, marginal discolouration, secondary caries, anatomical form, retention, postoperative sensitivity and colour matching. Restorations with an "Alpha (A)" score were considered successful, those with a "Bravo (B)" score were considered acceptable, and those with a "Charlie (C)" score were considered unsuccessful. The scoring of the restorations was decided by agreement of both dentists (Ryge G. et al., 1980).
The Schiff Cold Air Sensitivity Score | 1.5-2 year
  The Schiff Cold Air Sensitivity Score is a test conducted in dental units. Cold air from a spray is applied to the surface of the tooth's dentin, 2-3 mm away, and at a 90-degree angle, with continuous pressure of 45-60 PSI for 2-3 seconds, following the isolation of neighboring teeth. The temperature should be around 20 degrees Celsius. The patient's pain level is then scored by the dentist using a scale.
  * Score 0: No response to the stimulus.
  * Score 1: Responds to the stimulus but does not request it to be stopped.
  * Score 2: Responds to the stimulus, requests it to be stopped, or makes movements to avoid it.
  * Score 3: Responds to the stimulus, finds it painful, and requests it to be stopped.